CLINICAL TRIAL: NCT05005208
Title: SocIal ROBOTics for Active and Healthy Ageing
Acronym: SI-ROBOTICS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto Nazionale di Ricovero e Cura per Anziani (Other)
Collaborators: Ministero dell'Università e della Ricerca, Italia (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: INRCA_001_2021
Record Dates: First submitted 2021-08-05; First posted 2021-08-13 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Parkinson Disease; Aging
Keywords: Parkinson disease; Older people; Robot; Technology-integrated intervention; Rehabilitation
MeSH Terms: conditions — Parkinson Disease | interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rehabilitation Group (Experimental): PD subjects will be going through a rehabilitation program based on an Irish dance with the support of the technological platform SI-ROBOTICS
  Interventions: Other: rehabilitation program with the support of the technological platform SI-ROBOTICS

INTERVENTIONS:
Other: rehabilitation program with the support of the technological platform SI-ROBOTICS — A 16-treatment session will be conducted, divided into 2 training sessions per week, for 8 weeks. The therapy sessions last 60 minutes; each session will involve 2 patients at time. Cardiac and respiratory activity monitoring is planned during robotic treatments in order to detect the heart rate during physical activity. Individual participants must complete at least 80% of the sessions. Recovery of 2 sessions will be possible.
  Each session involves the following activities:
  * Breathing, relaxation and postural harmonization exercises;
  * Active mobility and stretching exercises;
  * Irish dance with the SI-ROBOTICS system;
  * Relaxation exercises.
  Other Names: SI-ROBOTICS a technological system facilitating a rehabilitation program

SUMMARY:
The study was designed to test the acceptability of the Si-Robotics system in a group of 20 subjects with Parkinson's Disease at an early stage, during a rehabilitation treatment based on Irish dancing. Assessments will be performed at the baseline and at the end of the treatment.

DETAILED DESCRIPTION:
The study was designed to test the acceptability of the SI-ROBOTICS system in a group of 20 subjects with Parkinson's Disease at an early stage during a rehabilitation treatment.

The SI-ROBOTICS system is composed of multiple technological components with the aim of facilitating a rehabilitation program based on Irish dance and encouraging the execution of dance steps. The SI-ROBOTICS system consists of:

* ROBOTIC PLATFORM: a social robot that allows the monitoring of patients during sessions, moving around patients safely and, if necessary, intervening in their support.
* LET'S DANCE GAME: a component that allows users to enjoy the game sessions (setting up of therapy sessions by the therapist, presentation of tasks to the player and execution by the latter, display of feedback on the sessions).
* ENVIRONMENTAL AND WEARABLE SENSORS: this allows data to be collected on the patient's main clinical parameters (e.g. heart rate, respiratory rate, etc.). These data allow the therapist to know the patient's state during the execution of tasks and the AI reasoner component to have an additional level of information with which to adapt the planning of steps.
* AI REASONERS: this is the back-end of the Si-Robotics system, i.e. the "intelligent" component that allows the adaptation of the game sessions, based on the users' game performance and the data collected through the sensors. In this way it will be possible to dynamically customize the session according to the user's needs and abilities.
* ARTIFICIAL VISION SETTING: a commercial camera called Inter Real Sense (https://www.intel.it/content/www/it/it/architecture-and-technology/realsense-overview.html) will be installed in the experimental setting for the extraction of kinematic parameters, saved anonymously and locally on this computer. Also the robotic platform will be equipped with a RealSense camera and will be able to acquire kinematic parameters. To extract features of interest from the signals, proprietary skeleton tracking software of the Real Sense camera will be used, together with specially developed algorithms for feature extraction.

In addition, kinematic and performance parameters will be collected, which will be used by the physiotherapist to evaluate and plan subsequent sessions, and by the system to delineate the levels of difficulty of the exercise.

ELIGIBILITY:
Inclusion Criteria:

* Capacity to consent;
* Hoen and Yahr scale: 1-2 stage;
* Functional Ambulation Category (FAC) ≥ 2;
* Ranking scale score ≤ 3;
* Stability of drug treatment for at least 1 month;
* Geriatric Depression Scale 4-items ≤ 1;
* Mini Mental State Examination ≥ 24;
* Maintaining an upright posture ≥ 30''.

Exclusion Criteria:

* History of syncopal episodes, epilepsy and vertigo not controlled pharmacologically;
* Serious dysfunction of the autonomic system;
* Severe behavioral syndromes not compensated by drugs;
* Concurrent neurological and/or cardiac diseases;
* Recent femur fracture
* Chronic medium to severe pain affecting standing or walking.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-05-19 (Actual); Primary Completion 2024-03-29 (Estimated); Study Completion 2024-03-29 (Estimated)

PRIMARY OUTCOMES:
Change in acceptability of the SI-ROBOTICS system | change from baseline to 4 and 8 weeks after intervention commencement
  Acceptability will be assessed using a 52-item questionnaire based on the unified theory of acceptance and use of technology (UTAUT) model. It's a standardized instrument for measuring the likelihood of success for new technology introductions and helps to understand the drivers of its acceptance.
  The questionnaire has 52 questions distributed in 4 key constructs: 1) performance expectancy, 2) effort expectancy, 3) social influence, and 4) facilitating conditions.
  Each question are based on a Likert-type 5-point scale ranging from 1 = strongly disagree to 5 = strongly agree. Increments are integers between 1 to 5.

SECONDARY OUTCOMES:
Change in walking speed | change from baseline to 4 and 8 weeks after intervention commencement
  The walking speed will be evaluated by the Six-Minute Walking Test (6MWT).
Change in balance | change from baseline to 4 and 8 weeks after intervention commencement
  The change in balance will be evaluated by the Performance-Oriented Mobility Assessment (POMA) consists of two sub-scales: the balance evaluation scale ("balance scale" or POMA-B) and the gait evaluation scale ("gait scale" or POMA-G). The maximum score is 28 points: in detail, the maximum score of the POMA-B is 16, while for the POMA-G the maximum score is 12.
Change in fear of falling | change from baseline to 4 and 8 weeks after intervention commencement
  The change in fear of falling will be evaluated by the Short Falls Efficacy Scale - International (FES-I- Short). The cut offs are divided as follows: a score between 7-8 indicates a low concern, between 9-12 a moderate concern and between 14 and 28, high concern.
Change in physical performance | change from baseline to 4 and 8 weeks after intervention commencement
  Change in physical performance will be ascertained using the Short Physical Performance Battery (SPPB). Summary scores range from 0-12 and higher scores denote higher physical performance
Change in mobility | change from baseline to 4 and 8 weeks after intervention commencement
  Change in mobility will be evaluated by Timed-Up-and-Go (TUG) Test. A score of ten seconds or less indicates normal mobility; times between 11 and 20 seconds are within normal limits for frail elderly and disabled patients; times over 20 seconds indicate that the person requires external assistance and the need for further examination and intervention. A score above 30 seconds suggests that the person may be prone to falls.
Change in goal attainment scale | change from baseline to 4 and 8 weeks after intervention commencement
  Change in goal attainment scale (GAS): definition of an individual goal at start, followed by a 6- point numeric scale indicating to what extent the goal is (score 0 till +2) or is not (-3 indicating detoriation till -1) reached.
Change in quality of life | change from baseline to 4 and 8 weeks after intervention commencement
  SF-12 Health Survey (SF-12) is composed of 12 items that produce two measurements related to two different aspects of health: physical health and mental health.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Riccardi, MD, Principal Investigator — IRCCS-INRCA
Locations (1):
- IRCCS INRCA Hospital, Ancona, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available to other researchers following a documented request to the INRCA investigators.

REFERENCES:
- [Derived] Bevilacqua R, Benadduci M, Bonfigli AR, Riccardi GR, Melone G, La Forgia A, Macchiarulo N, Rossetti L, Marzorati M, Rizzo G, Di Bitonto P, Potenza A, Fiorini L, Cortellessa Loizzo FG, La Viola C, Cavallo F, Leone A, Rescio G, Caroppo A, Manni A, Cesta A, Cortellessa G, Fracasso F, Orlandini A, Umbrico A, Rossi L, Maranesi E. Dancing With Parkinson's Disease: The SI-ROBOTICS Study Protocol. Front Public Health. 2021 Dec 21;9:780098. doi: 10.3389/fpubh.2021.780098. eCollection 2021. PMID 34993171